CLINICAL TRIAL: NCT04394403
Title: Pilot Internet-based Self-Help Program for Managing Corona Stress vs. Waitlist Control
Brief Title: Pilot Internet-based Self-Help Program for Managing Corona (COVID-19) Stress
Acronym: CoronaStress
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebrew University of Jerusalem (Other)
Responsible Party: Principal Investigator, Jonathan D. Huppert, Professor, Hebrew University of Jerusalem
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: coronastress
Record Dates: First submitted 2020-05-13; First posted 2020-05-19 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Stress; Stress, Psychological
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: This is a randomized trial to either immediate or delayed access to the internet guided self-help program
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immediate guided self-help (Experimental): In this condition, individuals will be given access to material and exercises based on CBT to reduce their stress
  Interventions: Behavioral: Internet-based guided self-help based on CBT principles
- waitlist (No Intervention): Individuals in this condition will wait 6 weeks before they are provided access to the guided self-help program

INTERVENTIONS:
Behavioral: Internet-based guided self-help based on CBT principles — Individuals are provided basic rationale of CBT to deal with stress, worry, anxiety, dysphoria, sleep difficulties, emotion dysregulation, and memories all related to COVID-19
  Other Names: ICBT for CoronaStress
  Arms: immediate guided self-help

SUMMARY:
The current study examines an adapted guided self-help stress reduction program, focusing on reducing stress in the time of COVID-19. Two studies are planned: 1) an international study in English in which individuals proficient in English throughout the world will participate and 2) a follow-up study in Hebrew.

DETAILED DESCRIPTION:
The current study examines an adapted guided self-help stress reduction program, focusing on reducing stress in the time of COVID-19. Two studies are proposed: 1) an international study in English in which individuals proficient in English throughout the world will participate and 2) a study in Hebrew. The first study will publicize via social media and participants will be randomized to either immediate participation or a 6 week waitlist period. Assessments will be conducted pre, (again after waitlist for the control group), posttx (after completion/cessation of the program), 6 month and 1 year followup. Two forms of assessment will be conducted: pre-post-follow-up (with the CRISIS measure) and weekly during the program (via the DASS-21). For the full program see: https://www.iterapi.se/sites/coronastress/

ELIGIBILITY:
Inclusion Criteria:

* Read/Write English,
* feels stress due to Corona/COVID-19

Exclusion Criteria:

* current psychological or psychiatric treatment,
* current psychiatric illness,
* suicidality,
* psychosis,
* bipolar,
* severe dissociative symptoms,
* in a currently severe traumatic situation,
* having a serious medical illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-05-14 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
The CoRonavIruS Health Impact Survey (CRISIS) | change from Pre to post treatment (6 weeks),
  change in a self-report measure of stress during the COVID-19 pandemic that ranges from 0-128. Higher means more symptomatic.
The CoRonavIruS Health Impact Survey (CRISIS) | change from Pre to 6 months Follow-up
  change in a self-report measure of stress during the COVID-19 pandemic that ranges from 0-128. Higher means more symptomatic.
The CoRonavIruS Health Impact Survey (CRISIS) | change from Pre to 1 year Follow-up
  change in a self-report measure of stress during the COVID-19 pandemic that ranges from 0-128. Higher means more symptomatic.

SECONDARY OUTCOMES:
Depression, Anxiety, and Stress Scale- 21 item version: DASS-21 | Weekly change during treatment and at pre and post (6 week) treatment evaluations
  a self-report measure of depression, anxiety and stress, with each subscale ranging from 0-28. Higher means more symptomatic.
Depression, Anxiety, and Stress Scale- 21 item version: DASS-21 | change from pre to 6 month follow up
  a self-report measure of depression, anxiety and stress, with each subscale ranging from 0-28. Higher means more symptomatic.
Depression, Anxiety, and Stress Scale- 21 item version: DASS-21 | change from pre to 1 year follow-up
  a self-report measure of depression, anxiety and stress, with each subscale ranging from 0-28. Higher means more symptomatic.

OTHER OUTCOMES:
completion rate of modules | 6 weeks
  how many modules each individual completes, with less than 2 being considered dropout

CONTACTS AND LOCATIONS:
Locations (1):
- Hebrew University of Jerusalem, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: site website for guided self-help program — https://www.iterapi.se/sites/coronastress/